CLINICAL TRIAL: NCT07329920
Title: Mesenchymal CTC Ratio Dynamics Predicts Response and Survival in Pancreatic Ductal Adenocarcinoma With Neoadjuvant/Conversion Therapy: a Large Single-center Retrospective Cohort Study
Brief Title: Mesenchymal CTC Ratio Dynamics Predicts Response and Survival in Pancreatic Ductal Adenocarcinoma With Neoadjuvant/Conversion Therapy
Status: Completed | Type: Observational
Sponsor: Guo ShiWei (Other)
Responsible Party: Sponsor-Investigator, Guo ShiWei, Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: Changhai Mesenchymal CTC R1
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Circulating Tumor Cells (CTCs); Neoadjuvant Therapy
Keywords: PDAC; Circulating tumor cells; Mesenchymal CTC ratio; Neoadjuvant therapy; Longitudinal detection; Cohort study
MeSH Terms: conditions — Neoplastic Cells, Circulating | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- none treatment group
- upfront surgery group
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- neoadjuvant/conversion therapy without surgery group
- neoadjuvant/conversion therapy with surgery group
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines

INTERVENTIONS:
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — Retrospective studies do not require intervention measures.
  Groups: neoadjuvant/conversion therapy with surgery group; upfront surgery group

SUMMARY:
The aim of this study was to evaluate the clinical utility of mesenchymal CTC ratio dynamics as a real-time biomarker for PDAC patients with neoadjuvant therapy.

DETAILED DESCRIPTION:
In this study, the investigators generated the largest PDAC patient cohort for CTC detection to date, which revealed mesenchymal CTC ratio dynamics as a robust biomarker during neoadjuvant therapy. The mesenchymal CTC ratio varied significantly across resectability status of PDAC with the highest level in the metastatic cohort. Moreover, the mesenchymal CTC ratio dynamics could be used for real-time assessment of neoadjuvant therapy response, accurate postoperative relapse surveillance and reliable prognostication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CTC detection at the time of PDAC diagnosis were collected from the prospective database. All patients were pathologically confirmed with PDAC by endoscopic ultrasound guided fine-needle aspiration or surgical resection specimens. According to therapeutic modalities, these patients were divided into four subgroups: none treatment group, upfront surgery group, neoadjuvant/conversion therapy without surgery group and neoadjuvant/conversion therapy with surgery group. All patients provided written informed consent to use their clinical data and samples.

Exclusion Criteria:

* Patients who could not tolerate neoadjuvant therapy or who had invasive intraductal papillary mucinous neoplasms, mucinous cystadenocarcinomas, or other non-pancreatic periampullary adenocarcinomas were excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent CTC detection at the time of PDAC diagnosis were collected from the prospective database. All patients were pathologically confirmed with PDAC by endoscopic ultrasound guided fine-needle aspiration or surgical resection specimens. According to therapeutic modalities, these patients were divided into four subgroups: none treatment group, upfront surgery group, neoadjuvant/conversion therapy without surgery group and neoadjuvant/conversion therapy with surgery group. All patients provided written informed consent to use their clinical data and samples.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Overall survival (OS) was defined as the interval from the date of diagnosis to the date of patient death or the last follow-up visit 1 month after surgery.

SECONDARY OUTCOMES:
Recurrence-free survival | Recurrence-free survival (RFS) was defined as the time interval from the date of diagnosis to the date of local or regional recurrence, distant metastases, death or the last follow-up visit 1 month after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobiliary and Pancreatic Surgery, First Affiliated Hospital of Naval Medical UniversityUniversity, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No